CLINICAL TRIAL: NCT03142048
Title: Community Intervention to Reduce Social Isolation in Elderly People in Disadvantaged Urban Areas: Study Protocol for a Mixed Methods Multi-approach Evaluation
Brief Title: Community Intervention to Reduce Social Isolation in Elderly People: a Mixed Methods Multi-approach Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Agency of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ES_2017
Record Dates: First submitted 2017-04-11; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-04

CONDITIONS: Social Isolation; Aging
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schools of Health for the Elderly (Experimental): Participants receiving the community intervention (explained in the section "Intervention")
  Interventions: Other: Schools of Health for the Elderly
- Comparison Group (No Intervention): Participants in the study that do not receive the intervention

INTERVENTIONS:
Other: Schools of Health for the Elderly — The intervention "School of Health for the Elderly " consists of 22 weekly group sessions of 1.5 hours each. In addition to helping participants learn about different health issues, the intervention encourages interaction among participants and works on personal skills. Furthermore, most sessions are led by professionals who are experts on the topic covered and work in the neighborhood (professionals from the health services, social services, markets or neighborhood associations), making it easier to inform participants of the neighborhood's available resources. The aim of the intervention is to decrease social isolation and loneliness and, therefore, to improve mental health, self-perceived health and wellbeing
  Arms: Schools of Health for the Elderly

SUMMARY:
Background:

The proportion of elderly people has dramatically increased in recent decades. Moreover, social and demographic trends show a global increase of elderly people at risk of loneliness and lack of social relationships. The objective of this study was to evaluate the process, the effectiveness and the cost-effectiveness of an intervention to reduce social isolation and its negative effects on health in elderly persons.

Methods:

This is a mixed methods multi-approach evaluation that includes: 1) A qualitative evaluation among coordinators and participants taking part in the intervention, through in depth-interviews and focus groups, respectively. The main topics covered will be positive and negative aspects of the intervention, suggestions for its improvement, opinions on different aspects of the intervention, and perceived benefits. 2) A quantitative quasi-experimental design, comparing a group of individuals taking part in the intervention with another group with similar characteristics not receiving the intervention. Data will be collected at the beginning and at the end of the intervention. Social support will be measured through questions drawn from the Medical Outcomes Study and the National Social Life, Health, and Aging Project questionnaires. Psychological morbidity will be measured through Goldberg's General Health Questionnaire, and Health-related Quality of Life will be measured through the EuroQoL questionnaire. Information on visits to the primary care center in the years before and after the intervention will be obtained from the electronic records of the primary care centers. 3) A cost-utility analysis, conducted from a health system (primary care) perspective, including direct costs of the program and the primary care health services used. The effects of the intervention will be measured on quality-adjusted life years.

Discussion:

There is an urgent need for studies assessing the effectiveness and the efficiency of potential interventions to reduce social isolation among elderly persons. The results of this study will help to fill the knowledge gap in this area and might be especially useful for the development of social and public health policies and programs for older people in disadvantaged neighborhoods in urban areas.

DETAILED DESCRIPTION:
Hypothesis:

The intervention evaluated in this protocol will significantly improve social support, mental health, general health status and distinct dimensions of quality of life in the intervention group (IG) compared with the comparison group (CG). Among participants in the IG, the intervention will also significantly reduce the number of visits to their primary care centers. Furthermore, this intervention will be cost effective.

Objectives:

General objective To evaluate the process, effectiveness and cost-effectiveness of an intervention to reduce social isolation and its consequent negative impact on health in the elderly.

Specific objectives

1. To evaluate the implementation process of the intervention (participant profile, positive and negative aspects of the intervention, barriers and facilitators in its implementation, quality of the intervention, and satisfaction).
2. To assess the impact of the intervention on social support, self-perceived health status, mental health and quality of life among participants, and visits to the primary care center.
3. To determine the cost-effectiveness of the intervention.

Methods:

Study design

This is a mixed methods multi-approach evaluation that includes:

* a qualitative evaluation among coordinators and participants who underwent the intervention through in-depth interviews and focus groups, respectively;
* a quantitative quasi-experimental design, comparing a group of individuals taking part in the intervention (IG) with another group with similar characteristics not receiving the intervention (CG). Data will be collected at the beginning and at the end of the intervention;
* an economic evaluation, which includes a cost-utility analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants signing the consent form

Exclusion Criteria:

* Participants with difficulties in maintaining participation for 6 months.
* Participants with difficulties in understanding or expressing themselves in Spanish or Catalan.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 135 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2015-09-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Psychological morbidity will be measured through Goldberg's General Health Questionnaire (GHQ | The outcome measure will be measured up to 12 months.
  The General Health Questionnaire (GHQ) is a psychometric screening tool to identify common psychiatric conditions.

SECONDARY OUTCOMES:
Visits to the primary care center will be measured through access to the electronic records of the primary care centers. | The outcome measure will be measured up to 12 months.
  Primary care centers have records of all the patient visits.
Health-related quality of life will be measured through the EuroQoL (EQ-5D) | The outcome measure will be measured up to 12 months.
  The EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
Social support will be also measured based on the "National Social Life, Health, and Aging Project" questionnaire | The outcome measure will be measured up to 12 months.
  The National Social Life, Health, and Aging project includes the measurement of social connectedness items
Social support based on Measures of Quality of Life Core Survey (MOS) | The outcome measure will be measured up to 12 months.
  The Medical Outcomes Study Social Support Survey cover four domains (emotional/informational support, tangible [also called instrumental] support, positive social interaction, and affection)

CONTACTS AND LOCATIONS:
Overall Officials: María José López, PhD, Principal Investigator — Public Health Agency of Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lapena C, Continente X, Sanchez Mascunano A, Mari dell'Olmo M, Lopez MJ. Effectiveness of a community intervention to reduce social isolation among older people in low-income neighbourhoods. Eur J Public Health. 2022 Oct 3;32(5):677-683. doi: 10.1093/eurpub/ckac100. PMID 36074028
- [Derived] Lopez MJ, Lapena C, Sanchez A, Continente X, Fernandez A; Evaluation Group of the "Schools of Health for older people". Community intervention to reduce social isolation in older adults in disadvantaged urban areas: study protocol for a mixed methods multi-approach evaluation. BMC Geriatr. 2019 Feb 18;19(1):44. doi: 10.1186/s12877-019-1055-9. PMID 30777022